CLINICAL TRIAL: NCT04300257
Title: Swiss Sarcoma Network: Prediction Model for Patient Selection in Sarcoma Care
Status: Recruiting | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Swiss Sarcoma Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-01107
Record Dates: First submitted 2020-02-20; First posted 2020-03-09 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sarcoma
Keywords: Sarcoma, Epithelioid; Sarcoma, Soft Tissue; Sarcoma, Spindle Cell; Sarcoma, Bone
MeSH Terms: conditions — Sarcoma; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary significance of this project is to perform a detailed analysis to assess the diagnostics, treatment and follow-up care, to develop a prediction model for future patient selection regarding various diagnostic and treatment procedures.

DETAILED DESCRIPTION:
Within the framework of interdisciplinary cooperation for a sarcoma problem, predictive and prognostic criteria will be developed that improve the treatment and particularly outcome.

The outcome variables include patient characteristics, tumor types and characteristics, histology, management and treatment strategies as well as recurrence rate and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Malignant and intermediate and selected benign bone or soft tissue tumors, acc. to the WHO coding list of the SSN
* Female and male subjects of all ages

Exclusion Criteria:

* Documented objection of subsequent use of personal health data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from bone or soft tissue tumors.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10-19 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis, | 5 years
  Data collected in the registry will be evaluated and analyzed to determine criteria to improve treatment strategies
Local recurrence, | 5 years
  s.o.
distant metastasis, | 5 years
  s.o.
biopsy taken by operating surgeon-radiologist-team, | 5 years
  s.o.
pathology centrally reviewed, | 5 years
  s.o.
Surgery (yes/no), | 5 years
  s.o.
Surgical margin status, | 5 years
  s.o.
surgery performed by dedicated surgeon, | 5 years
  s.o.
Radiation Therapy (yes/no), | 5 years
  s.o.
Chemotherapy (yes/no), | 5 years
  s.o.
decision of board carried out, | 5 years
  s.o.
Status at last contact, | 5 years
  s.o.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Fuchs, Prof, Principal Investigator — SwissSarcomaNetwork
Locations (8):
- Switzerland (8):
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - SwissSarcomaNetwork, Winterthur, Canton of Zurich
  - Ente Ospedaliero Cantonale, Bellinzona, Canton Ticino
  - Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Luzerner Kantonsspital, Lucerne
  - Pathologie Institut Enge, Zurich
  - Klinik Hirslanden, Zurich
  - Stadtspital Zürich Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andritsch E, Beishon M, Bielack S, Bonvalot S, Casali P, Crul M, Delgado Bolton R, Donati DM, Douis H, Haas R, Hogendoorn P, Kozhaeva O, Lavender V, Lovey J, Negrouk A, Pereira P, Roca P, de Lempdes GR, Saarto T, van Berck B, Vassal G, Wartenberg M, Yared W, Costa A, Naredi P. ECCO Essential Requirements for Quality Cancer Care: Soft Tissue Sarcoma in Adults and Bone Sarcoma. A critical review. Crit Rev Oncol Hematol. 2017 Feb;110:94-105. doi: 10.1016/j.critrevonc.2016.12.002. Epub 2016 Dec 8. PMID 28109409
- [Result] Abarca T, Gao Y, Monga V, Tanas MR, Milhem MM, Miller BJ. Improved survival for extremity soft tissue sarcoma treated in high-volume facilities. J Surg Oncol. 2018 Jun;117(7):1479-1486. doi: 10.1002/jso.25052. Epub 2018 Apr 6. PMID 29633281